CLINICAL TRIAL: NCT00412386
Title: Abnormal 3-dimensional MRI Flow Patterns and Plasma Matrix Metalloproteinase Levels Predict Dilatation of Ascending Aorta in Adolescent Patients With Bicuspid Aortic Valve
Brief Title: Abnormal 3-D MRI Flow Patterns in Adolescents Patients With Bicuspid Aortic Valve
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, Denver Sallee, Assistant Professor, Emory University
Other Study IDs: IRB00000134
Record Dates: First submitted 2006-12-14; First posted 2006-12-18 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-12

CONDITIONS: Congenital Heart Disease; Bicuspid Aortic Valve
Keywords: Pediatric; Congenital Heart Disease; Imaging
MeSH Terms: conditions — Heart Defects, Congenital; Bicuspid Aortic Valve Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- BAV: patients with BAV
- Normal control: normal patients

SUMMARY:
Bicuspid aortic valve (BAV) is a form of congenital heart disease (the person is born with it). With BAV, the heart valves in the aorta (the blood vessel that takes blood away from the heart to the body) are not formed right. A person with BAV has only 2 leaflets instead of three and the valve leaflets are often thickened. This can result in the block of blood flow across the valve (aortic stenosis) and/or valve leakage (aortic valve regurgitation).

From our experience at least 1/3 of patients with BAV will eventually develop complications. Many patients with BAV do not develop significant problems until well into adulthood. The most common problem in BAV patients is aortic dilatation and/or dissection. At this point, we do not know on who or why aortic dilatation or dissection occurs.It is unclear whether the enlargement is because of abnormal blood flow patterns, as a result of the shape of the bicuspid valve, or whether it is because the way the aortic valve and/or vessel is formed. In other words, the abnormal shape of the aortic valve may cause blood to flow in a different way than it normally would, causing damage to the aorta as blood leaves the heart. There may be a problem with the way the aortic valve connects to the aorta, which causes the aorta to get larger or break down over time. It is also possible that the wall of the aorta in patients with BAV is weaker than it would be in patients without BAV. At this point, we do not know. It is believed by the investigators that if we can determine why the aorta gets larger or tears, we can minimize the effects or prevent them altogether.

This study will collect blood and cardiac MRI images from forty-five (45) patients at Children's Healthcare of Atlanta Egleston. There will be a study group (patients with BAV) and a control group of patients (patients scheduled for a cardiac MRI but without BAV).

All enrolled patients will have blood drawn by nursing staff from a peripheral vein and collected in tubes for testing the day of their MRI scan. This test is called a plasma matrix metalloproteinase level. It is believed that patients who have bicuspid aortic valves and dilated aortas have high plasma levels of this protein. This study will compare the MRI images and plasma matrix protein levels of all the patients participating in the study.

DETAILED DESCRIPTION:
Introduction-Background The reported incidence of bicuspid aortic valve (BAV) based largely on autopsy studies varies between 0.4% to 2.25% of the population. At least a third of patients with a bicuspid aortic valve will eventually develop complications which include aortic stenosis, aortic regurgitation, infective endocarditis, aortic dilatation, aortic aneurysm formation, or aortic dissection. Given that in combination all other forms of congenital heart disease are thought to be present in 0.8% of live births, Ward has suggested that bicuspid aortic valves are likely to result in more morbidity and possibly mortality than the effects of all other congenital heart defects combined. Since many patients with bicuspid aortic valves do not develop significant problems until well into adulthood, clinicians have not focused much attention on the "normally" functioning bicuspid aortic valve. However, at a mean age of 17.8 years 52% of males with normally functioning aortic valves already have aortic dilatation, implying that associated aortic stenosis and/or regurgitation is not an obligate precursor.

Previous studies have demonstrated an association between bicuspid aortic valves and dilatation of the aorta. Gurvitz et al. performed echocardiographic measurements of the aortas of children and found that those with bicuspid aortic valves had significantly larger aortas compared with controls, regardless of the presence of aortic stenosis or regurgitation. Nevertheless, the definition of clinical predictors of the risk for the development of aortic dilatation/dissection and an understanding of the mechanisms leading to aortic dilatation are lacking. Specifically, it remains unclear as yet whether such dilatation is secondary to abnormal flow patterns and shear stresses resulting from the bicuspid valve morphology or whether it is a manifestation of a distinct underlying structural problem with not only the aortic valve but also the aortic root including the ascending aorta.

Fernandes et al. recently reviewed the echocardiograms of 1,135 children with bicuspid aortic valves and found that there were differences among the patients related to aortic valve morphology. For instance, associated moderate or greater aortic stenosis was present in 9.7% of patients with fusion of the intercoronary commissure of the aortic valve, vs 25.9% of patients with fusion of the right-coronary and non-coronary commissure, and in none of the patients with fusion of the left coronary and non-coronary aortic valve leaflets. Moreover, fusion of the right coronary and non-coronary cusps resulted in a two-fold higher risk of at least moderate aortic regurgitation compared with the other types of bicuspid aortic valves. However, this generalized division of bicuspid aortic valves into three types based on which commissure is fused is likely an oversimplification, and Fernandes did not report on the relationship between valve morphology and aortic root dilatation. However, Novaro et al. found that adult patients (mean age of 54 year) with fusion of the right/non-coronary commissure tended to have larger mid-ascending aortas compared with patients with fusion of the intercoronary commissure, but the difference did not reach statistical significance. Nevertheless, both personal clinical observations and recent publications support the assertion that individual bicuspid aortic valves may function quite differently from one another. For instance, there are bicuspid aortic valves in which there are two nearly symmetric leaflets whereas others may have a dominant cusp to varying degrees, resulting in a markedly eccentric orifice when the valve opens. In an elegant experimental model using excised bicuspid valves analyzed with intravascular ultrasound and high-resolution videography, Robicsek et al demonstrated that asymmetric bicuspid valves "induced extensive recirculation vortices in the ascending aorta." They found that the vortex was not "trapped" in the sinuses of Valsalva as it is in a normal tricuspid aortic valve, but instead is extended into the ascending aorta and aimed toward the right anterolateral aspect of the aorta (the convexity of the aorta). This correlates with published reports and our own personal experience in performing clinical cardiac magnetic resonance imaging (CMR) studies on patients with bicuspid aortic valves and aortic root dilatation in whom there is oft-noted asymmetry in the pattern of dilatation of the ascending aorta and resulting in an oval-shaped rather than a circular aortic root and ascending aorta.

Extrapolating from the studies of Robicsek, variations present in the geometry of bicuspid valves are likely to result in varying degrees of turbulence even in the absence aortic valve stenosis. In theory, the turbulent blood flow directed at a particular segment of the aortic wall may result in local changes to the aortic wall leading to asymmetric aortic dilatation. These changes are postulated to result from receptors present on both endothelial and smooth muscle cells that have the ability to adapt to sheer stress by altering local gene expression which in turn modulates the tension between focal adhesion sites, integrins, and the extracellular matrix. Moreover, fibrillin-1, which is deficient in patients with dilated aortic roots and Marfan syndrome, has also been found to be deficient in the aortas of patients with bicuspid aortic valves. Similarly, Cotrufo et al. found asymmetric patterns of matrix protein expression and content and asymmetric patterns of elastic medial wall degeneration in the aortic walls of patients with bicuspid aortic valves. In addition, these investigators found differences between patients with bicuspid aortic valves and associated stenosis vs regurgitation, suggesting that focally-directed aortic turbulence may be influencing local gene expression and potentially explaining the asymmetric pattern of aortic dilatation that is often observed. Lastly, several recent studies have highlighted the relationship between circulating plasma MMP-2 and MMP-9 levels either in aortic dilatation in adult patients with thoracic or abdominal aortic aneurysms or in adults with aortic dilatation secondary to systemic hypertension. In addition, histologic examination of aortic aneurysm tissue in adult patients with bicuspid aortic valves demonstrated increased MMP-2 expression vs. aortic aneurysms in adults with trileaflet aortic valves.

Recently investigators have used cardiac MRI (CMR) to study flow patterns in the aorta. CMR is a noninvasive technique that permits 3-dimensional anatomic characterization as well as assessment of aortic flow. Markl et al. have used time-resolved 3-dimensional phase-contrast magnetic resonance imaging (3D-PCMRI) techniques to characterize aortic flow in both normal adults and in adults after aortic root replacement. These authors established that 3-dimensional magnetic resonance velocity mapping was a useful technique to visualize and qualitatively assess the complex aortic flow patterns in both normal controls and in patients with aortic pathology. Similarly, Kvitting et al., who studied both adult volunteers and 2 patients with Marfan syndrome following aortic valve sparing operations, found that the alterations to the normal aortic sinus architecture following surgery resulted in a loss of the normal vortical flow patterns seen in the aortic sinuses.

Specific Aims

1. Develop clinically feasible MRI imaging strategies to perform a complete evaluation of structure and functional dynamics of the heart, including the aortic valve, aortic root, and ascending aorta, as well as full volumetric 3-D ciné flow velocity encoding of the entire aortic root region and proximal ascending aorta.
2. Define qualitative and quantitative metrics to characterize different types of bicuspid aortic valve morphology and flow patterns. These metrics will be based on structural information and the blood flow patterns in the aortic root, observed in MRI studies of patients with diagnosed bicuspid aortic valves, as compared to observation in control subjects with known normal aortic valves and anatomy of ascending aorta.
3. Correlate different bicuspid aortic valve morphologies and observed characteristic flow patterns with the risk of development of aortic dilatation at various levels of the aorta, such as the aortic root, proximal ascending aorta, and distal ascending aorta.
4. Quantify plasma concentrations of matrix metalloproteinase-2 (MMP-2) and matrix metalloproteinase-9 (MMP-9) levels as well as the levels of their specific tissue inhibitors, respectively tissue inhibitor of metalloproteinase-2 (TIMP-2) and tissue inhibitor of metalloproteinase-1 (TIMP-1) in controls and bicuspid aortic valve patients.
5. Correlate biochemical markers of extracellular matrix degradation (both MMP and TIMP) with the presence or absence of aortic dilatation in both controls and in patients with bicuspid aortic valves.

Study Design We will prospectively perform cardiac magnetic resonance studies on 30 patients, ages 10-18 years with known bicuspid aortic valves (BAV), and on 15 normal control subjects. The BAV patient population will consist of 15 patients with aortic root dilatation for body surface area as determined by published pediatric echocardiographic normal values and 15 without aortic dilatation. Echocardiographic normals indexed for body surface area will be used, as there are no published normal CMR values for aortic dimensions in pediatric patients using cine MR techniques; however aortic measurements by echocardiography and CMR in a pediatric patient population have been shown to reveal no significant differences except for the descending aorta. Since either significant aortic stenosis or regurgitation has been associated with aortic dilatation, patients will be excluded if they have more than mild stenosis or regurgitation.

As in previous published reports, mild aortic stenosis will be classified as a mean gradient across the aortic valve <17 mmHg on routine clinical echocardiography. Mild aortic regurgitation will be defined on routine clinical echocardiography as resulting in a left ventricular end-diastolic dimension <2 standard deviations below the mean for body surface area and the absence of pan-diastolic retrograde flow on pulsed Doppler evaluation of the abdominal descending aorta. Studies will be performed without sedation, but with breath-holding instructions as appropriate.

Controls will consist of 15 patients with normal aortic valves and aortas who are undergoing clinically indicated CMR studies for reasons such as chest pain or assessment for cardiomyopathy and who are found to have structurally/functionally normal hearts.

MRI Methods Cardiac magnetic resonance (CMR) studies will be performed in a GE 1.5 T MR system with Release 12M4 cardiovascular software. MR imaging will focus on of visualization in high definition of the anatomy of the aortic valve and aortic root utilizing 2-dimensional and 3-dimensional FIESTA cine MR sequences. Flow data will be acquired using 2-dimensional, or, whenever allowed within imaging time constraints, fully 3-dimensional phase velocity mapping sequences with full vector-encoding of velocities at 200 cm/s maximum velocity encoding VENC, adjusted up if velocity aliasing is observed. For 2-D flow acquisitions in planes across the main flow direction the in-plane directional components may be acquired at lower velocity encoding to achieve higher accuracy. To resolve blood flow and cardiovascular anatomy as a function of the cardiac phase (cine imaging), image acquisition will be synchronized with the vector cardiogram to reconstruct approximately 16-20 cine images representing the different phases of the cardiac cycle. Initial data acquisition for structural and velocity-encoded imaging will be performed with standard pulse sequence software as supplied by General Electric with the imaging device. These scans will initially be acquired in free-breathing mode. A series of 5-10 studies on normal volunteers will be conducted to optimize the protocol within those constraints, and develop guidelines for an prescribed add-on imaging protocol, ideally limited to not more than 20 minutes of scan time, for acquisition of the aortic scans. Priority solutions for respiratory motion compensation during the acquisition depending on the demonstrated reliability of the available options (free-breathing, breath-holding, respiratory k-space ordering, navigator- or belt & bellows-monitored respiratory gating) in these volunteer test studies, and based on the capability of each study subject to accommodate these options. The scans defined in this protocol will be added initially to the clinical protocol of all subjects in the study. In parallel with the protocol development and implementation by standards pulse sequence methods, we will pursue a collaboration effort with the MRI imaging resource center at Stanford University. The Stanford group has developed a highly optimized image acquisition method which allows fully vector-encoded 3-D respiration-ordered acquisition of an arbitrarily positioned rectangular 3-D imaging volume. We anticipate that this acquisition software, which will require running specialized pulse sequence software and off-line image reconstruction on one of our computer workstations, will improve the coverage and overall resolution of the flow-encoded data significantly. We have the required expertise and research software tools available from General Electric, but currently only enabled for research on the WCI scanner at Emory. For this project, but possibly concurrently with transition of software development efforts for other research projects (Noquist project) we will request authorization from GE to run the required research patches on the Egleston 1.5T GE instrument.

Plasma MMP and TIMP quantification methods Blood samples will be taken from peripheral veins by nursing staff.MMP and TIMP levels will then be measured using commercially available sandwich enzyme-linked immunosorbent assay (ELISA) kits which have previously been validated for use in human tissue homogenates.Serum MMP levels will be determined using MMP-2 and MMP-9 monoclonal antibodies.Levels of TIMP-1 and -2 will be determined using monoclonal antibodies.

Image Processing Methods Visualization and quantitative analysis of velocity mapping data will be performed, initially exclusively, utilizing in-house HeartViz software developed by Marijn Brummer, Ph.D.The current version of the software allows fully interactive 3-D dynamic integrated display of structural information through texture-mapped slice display and time-resolved volume rendering, in conjunction with dynamic flow vector field visualization from multiple flow acquisitions in the same view. This software has been developed by the investigators during the past ten years, and has been proposed and used for evaluation of a variety of congenital and acquired cardiac diseases, including aortic coarctations, VSD, aortic dissections, and peri-atrial tumors.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with Bicuspid Aortic Valve 15 with aortic root dilatation 15 without aortic root dilatation
* 15 patients with congenital heart disease, but not bicuspid aortic valve
* meet eligibility criteria for MRI
* 10-18 years of age

Exclusion Criteria:

* under 10 years and over 19 years of age
* systemic hypertension for age and height
* Marfan syndrome
* on cardiac or vasoactive medications
* contra-indications to MRI such as metallic implants
* acquired heart disease
* require sedation

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: patients with bicuspid Aortic valve, normal healthy volunteers, and congential heart disease without bicuspid aortic valve
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2006-12; Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denver Sallee, MD, Principal Investigator — Emory University
Locations (1):
- Childrens Healthcare of Atlanta, Atlanta, Georgia, United States

REFERENCES:
- [Background] Robicsek F, Thubrikar MJ, Cook JW, Fowler B. The congenitally bicuspid aortic valve: how does it function? Why does it fail? Ann Thorac Surg. 2004 Jan;77(1):177-85. doi: 10.1016/s0003-4975(03)01249-9. PMID 14726058
- [Background] Fernandes SM, Sanders SP, Khairy P, Jenkins KJ, Gauvreau K, Lang P, Simonds H, Colan SD. Morphology of bicuspid aortic valve in children and adolescents. J Am Coll Cardiol. 2004 Oct 19;44(8):1648-51. doi: 10.1016/j.jacc.2004.05.063. PMID 15489098
- [Background] Novaro GM, Tiong IY, Pearce GL, Grimm RA, Smedira N, Griffin BP. Features and predictors of ascending aortic dilatation in association with a congenital bicuspid aortic valve. Am J Cardiol. 2003 Jul 1;92(1):99-101. doi: 10.1016/s0002-9149(03)00480-6. No abstract available. PMID 12842261
- [Background] Karakaya O, Barutcu I, Esen AM, Dogan S, Saglam M, Karapinar H, Akgun T, Karavelioglu Y, Esen O, Ozdemir N, Turkmen S, Kaymaz C. Relationship between circulating plasma matrix metalloproteinase-9 (gelatinase-B) concentration and aortic root dilatation. Am J Hypertens. 2006 Apr;19(4):361-5. doi: 10.1016/j.amjhyper.2005.08.013. PMID 16580570